CLINICAL TRIAL: NCT03389594
Title: Assesment of the Accuracy of Surgical Guide Designed From CBCT With Different Voxel Size in Computer Guided Implantology Randomized Clinical Trial
Brief Title: Assesment of the Accuracy of Surgical Guide Designed From CBCT With Different Voxel Sizes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Mohammed Ahmed Elhag, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ElhagCUImplant
Record Dates: First submitted 2017-12-13; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Accuracy of Surgical Guide in Implants
Keywords: Surgical guide; Computer guided implantology; CBCT voxel size

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each patient will be given a code by researcher (M.H) and the observers will be blind to which group this case belong
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical guide designed from voxel size 0.2mm (No Intervention): Surgical guide will be designed based on CBCT voxel size 0.2mm
- Surgical guide designed from voxel size 0.4m (Active Comparator): Surgical guide will be designed based on CBCT voxel size 0.4 mm
  Interventions: Other: Surgical guide

INTERVENTIONS:
Other: Surgical guide — Surgical Guide for this group will designed from 0.4mm voxel size
  Arms: Surgical guide designed from voxel size 0.4m

SUMMARY:
Accuracy Of CBCT affected by many factors. On of the most factors the affect the image quality is voxel size. Larger voxel size give a higher accuracy of the images but with higher radiation dose.

The study is to assist the accuracy of surgical guides designed from CBCT with different voxel sizes .

DETAILED DESCRIPTION:
Accuracy Of CBCT affected by many factors. On of the most factors the affect the image quality is voxel size. Larger voxel size give a higher accuracy of the images but with higher radiation dose.

The study is to assist the accuracy of surgical guides designed from CBCT with different voxel sizes (voxel size 0.4mm & 0.2mm)

ELIGIBILITY:
Inclusion Criteria:

* partially edentulous patients seeking for dental implant
* Bucco-lingual width more than 6 mm
* Medically free patients

Exclusion Criteria:

* patients with thin ridges that may need augmentation
* patients with systematic diseases that may affect bone quality
* completely edentulous patients
* patients with limited mouth opening

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-15 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Angular deviation | Immediate post operative
  Evaluation of angular deviation of virtual implant and actual implant positions according to voxel size difference (0.2 mm versus 0.4 mm)
Linear deviation | Immediate post operative
  Evaluation of linear deviation of virtual implant and actual implant positions according to voxel size difference (0.2 mm versus 0.4 mm

CONTACTS AND LOCATIONS:
Overall Officials: Cairo university, Principal Investigator — Cairo University, Faculty of dentistry
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided